CLINICAL TRIAL: NCT07049159
Title: A Two-stage, Phase 2b, Randomized, Double-blind, Placebo-controlled Safety, and Efficacy Study of ShigETEC, a Live, Attenuated, Oral Combination Vaccine to Prevent Shigella and ETEC Disease Delivered to Healthy Adults Ages 18 to 50 Years Old
Brief Title: Safety, and Efficacy Study of ShigETEC, a Live, Attenuated, Oral Combination Vaccine to Prevent Shigella and ETEC Disease Delivered to Healthy Adults Ages 18 to 50 Years Old
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eveliqure Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EVQ2001 / DMID 23-0009
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Shigella
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ShigETEC, a live, attenuated, oral vaccine (Experimental): Eligible participants will be randomly assigned in a 1:1 ratio to receive either ShigETEC 5x10^10 colony forming units (CFU) or placebo. Participants will receive their assigned treatment on Days 1, 4, 7, and 10.
  Interventions: Biological: ShigETEC vaccine; Biological: Challenge: Shigella flexneri 2457T at a dose of 1.5x10^3 CFU
- Placebo (Placebo Comparator): Eligible participants will be randomly assigned in a 1:1 ratio to receive either ShigETEC 5x10^10 colony forming units (CFU) or placebo. Participants will receive their assigned treatment on Days 1, 4, 7, and 10.
  Interventions: Other: Placebo; Biological: Challenge: Shigella flexneri 2457T at a dose of 1.5x10^3 CFU

INTERVENTIONS:
Biological: ShigETEC vaccine — The ShigETEC vaccine will be administered orally 4 times at 3-day intervals as a bacterial suspension in a volume of 30 mL per dose (target to contain 5x10^10 CFU)
  Arms: ShigETEC, a live, attenuated, oral vaccine
Other: Placebo — Eligible participants will be randomly assigned in a 1:1 ratio to receive either ShigETEC 5x10^10 colony forming units (CFU) or placebo. Participants will receive their assigned treatment on Days 1, 4, 7, and 10.
  Arms: Placebo
Biological: Challenge: Shigella flexneri 2457T at a dose of 1.5x10^3 CFU — In the challenge stage all participants will receive 1 oral dose of Shigella flexneri 2457T at a dose of 1.5x10^3 CFU.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the oral, live, attenuated ShigETEC vaccine against challenge with S. flexneri 2457T.

In Stage 1 of this study, ShigETEC vaccine or placebo will be administered orally to healthy participants at a dose of 5x10^10 CFU. This dose was tested in a Phase 1 trial and found to be safe when given 4 times with an interval of 3 days between each dose.

The efficacy of ShigETEC vaccination will be evaluated in Stage 2 of this study, when participants will be challenged with S. flexneri 2457T.

The study population will be healthy adult participants in the age of 18-50 years (inclusive), which are clearly defined in the study protocol.

DETAILED DESCRIPTION:
This is a two-stage, randomized, double blind, placebo-controlled Phase 2b study in healthy participants conducted at a single site.

The study will be conducted in two Stages (Stage 1 and Stage 2) and two arms in Stage 1 (Arm 1 and Arm 2).

Stage 1 Stage 1 will be conducted in an outpatient setting and includes the vaccination with the investigational product, ShigETEC, a live, attenuated, oral vaccine (Arm 1) and placebo (Arm 2) and subsequent follow-up.

Stage 2 Stage 2 will include an infectious challenge of selected Stage 1 participants in an inpatient setting (CHIM: Controlled Human Infection Model) in which participants will receive 1 oral dose of Shigella flexneri 2a 2457T and be followed closely for the signs and symptoms of shigellosis.

Stage 2 will start 21 (+5) days after the last dose of vaccine or placebo.

ELIGIBILITY:
Inclusion Criteria for stage 1:

1. Generally healthy non-pregnant, non-nursing adults aged 18 to 50 years.
2. Who are determined by medical history, physical examination, laboratory testing, and clinical judgment to be eligible for this study.
3. Who provide written informed consent after the nature of the study had been explained.
4. Who are available for the duration of the trial (from enrollment to study completion).
5. Who are able to understand and are willing to comply with all study requirements, and willing to follow the instructions of the study staff and complete a comprehension test.
6. Who have a body mass index (BMI) ≥19 and <40 kg/m2.
7. Participants of child-bearing potential must agree to avoid pregnancy throughout the study until 29 days following the challenge dose by use of an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable if it is a lifestyle choice (not just to participate in the study). If the participant is abstinent at the time of signing the informed consent and becomes sexually active, they must agree to use contraception as described. Participants who are unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).
8. Who are willing to not smoking during inpatient stay.
9. Who are willing to refrain from participating in other studies of investigational products until completion of the last study visit.

Exclusion Criteria for stage 1:

1. Participants who are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period.
2. Presence of a significant medical or psychiatric condition which in the opinion of the Investigator precludes participation in the study.
3. Clinically significant abnormalities in screening hematology or serum chemistry, defined as > grade 1 abnormality of serum potassium, alanine aminotransferase (ALT) or creatinine, hemoglobin, white blood cell count (WBC), or neutrophil count.
4. Who have received any blood products, including immunoglobulin, in the period from 6 months prior to vaccination or are anticipated to receive such products through to the conclusion of the study and have not donated blood within 30 days and agree not to donate blood until 1 year after challenge.
5. Who are receiving systemic antibiotics, completed antibiotic therapy, or receiving probiotics, prebiotics or synbiotics in previous 7 days before vaccination, or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing with vaccine.
6. Who have an immunosuppressive condition or IgA deficiency (serum IgA <7 mg/dl or limit of detection of assay) or evidence of impaired immune function, either congenital, acquired, or iatrogenic.
7. Who have or are participating in or have concluded participation in a clinical research study in the last 30 days or have not cleared the experimental product prior to vaccination.
8. Received a live vaccine within 30 days before scheduled receipt of IP; or an inactivated vaccine within 14 days before scheduled receipt of IP.
9. Who have a chronic non-gastrointestinal medical condition (e.g., hypertension, hyperlipidemia) that is not well controlled with medication.
10. Who have a significant history of or current diagnosis of diseases of the gastrointestinal tract (i.e., liver, gallbladder, bowel, or stomach), including inflammatory bowel disease, are on medication for such disease, or have had significant bowel surgery (with the exclusion of hernia repair, cholecystectomy, or appendectomy).
11. Presence of HIV antibody, HBsAg, or HCV antibody (if confirmed positive by HepC confirmatory test, i.e., recombinant immunoblot assay, PCR).
12. Who have a personal or family history of reactive arthritis or are HLA B-27 positive and therefore at risk for developing reactive arthritis following naturally acquired bacterial gastrointestinal infection.
13. Who work as a food handler or in direct patient, child day care, or elder care.
14. Who have immunocompromised household member.
15. Who have a child under the age of 2 living in their household.
16. Who have had a culture proven Shigella or ETEC infection within the last 5 years.
17. Who have a serum IgG titer >2500 to Shigella flexneri 2a.
18. Who have regularly abnormal stool patterns (fewer than 3 stools per week or more than 3 stools per day) or loose or liquid stools.
19. Who regularly use antidiarrheals, laxatives or any agents modulating gastric pH (regular defined as at least weekly).
20. Who have known allergy to 2 of the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole or ampicillin.
21. Who have known intolerance or allergy against polyethylene glycol (PEG); or corn starch.
22. Who have known intolerance or allergy to soy.
23. Who have personal history of or first-degree family member with an autoimmune disease.
24. Use any medication known to affect the immune function (e.g., systemic steroids) within 30 days preceding the first vaccination or planned use during the entire study period.
25. Who received an investigational or licensed vaccine against shigella, cholera, ETEC and/or LT toxin.
26. Who are dependent of the Sponsor, of the investigational team or his/her immediate family or are students of the professors at the clinical study site.
27. Who have evidence of current excessive alcohol consumption or drug dependence.
28. Current occupation involving handling of Shigella and ETEC bacteria.
29. Any other criteria which, in the Investigator's opinion, would compromise the ability of the participant to participate in the study, the safety of the study, or the results of the study.

Inclusion / Exclusion criteria for challenge

Only participants meeting the above inclusion/exclusion criteria and the additional following criteria at Stage 2 study entry are eligible to be in Stage 2:

1. Who received 4 doses of vaccine or placebo.
2. Who are SARS-COV-2 negative.
3. Who do not have an ongoing grade 2 or higher AE.
4. Who have negative pregnancy test (participants with child-bearing potential).
5. Who have not experienced diarrhea in the 7 days before challenge.
6. Who have not taken antibiotics, probiotics, prebiotics or synbiotics in the previous 7 days before challenge.
7. Who did not use anti-diarrheal, anti-constipation drugs within 7 days before challenge.
8. Who did not use proton pump inhibitors, H2 blockers or antacid therapy 48 hours prior to challenge.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the ShigETEC vaccine in preventing shigellosis caused by the challenge strain | Up to study day 60
  The proportion of participants with incidence of shigellosis caused by the challenge strain in vaccine vs. placebo recipients until the start of antibiotic administration.

SECONDARY OUTCOMES:
Safety and tolerability of ShigETEC oral vaccine | Up to 12 months after last vaccination
  * Number and severity of gastrointestinal and other solicited symptoms (specified as reactogenicity events) up to Day 16 (6 days after last vaccination)
  * Number and severity of unsolicited AEs up to Day 60 (28 days after challenge)
  * Number and severity of SAEs/MAAEs/pIMD up to Day 375 (12 months after last vaccination)
  * Number and severity of AEs of special interest
Characterization of the challenge strain shedding in stool samples | Up to study day 40
  Number and percentage of participants with detectable presence of challenge strain in stool samples detected by quantitative or qualitative culture or polymerase chain reaction (PCR).
Severity of disease following challenge using Shigella disease score | Up to day 40
  Maximum disease severity following challenge in the vaccinated vs placebo groups using the Shigella disease score.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Immunization Research, Baltimore, Maryland, United States